CLINICAL TRIAL: NCT06090201
Title: Cerebral Microbleeds in Severe Congenital Hemostatic Defects: Prevalence and Impact on Cognition
Brief Title: Severe Congenital Hemostatic Defects, Cerebral MIcrobleeds and COGnition
Acronym: HEMICOG
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_0601
Record Dates: First submitted 2023-10-05; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Microbleeds, Congenital Haemophilia, Congenital Von Willebrand Disease
Keywords: Cerebral microbleeds (CMBs); Congenital haemophilia; Congenital von Willebrand disease (vWd); Cerebral small vessel disease (SVD); Cognition; Magnetic resonance imaging (MRI)
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 3-Tesla brain MRI and a comprehensive neuropsychological assessment — Patients with a moderate to severe form of congenital haemophilia A or B or a severe form of von Willebrand disease will be consecutively recruited in the study during a routine follow-up visit at the Haemostasis and Transfusion Department of the Lille University Hospital.

SUMMARY:
Cerebral microbleeds (CMBs) are haemosiderin deposits, resulting from the leakage of erythrocytes from small cerebral vessels, which can be detected noninvasively using susceptibility-sensitive magnetic resonance imaging (MRI) techniques. CMBs are commonly observed in daily practice: their prevalence range from five percent in healthy individuals over 65 years old to 50% in patients with a history of stroke. CMBs are associated with intracerebral hemorrhage (ICH) and also cognitive impairment and dementia.

The pathophysiology of CMBs is thought to primarily involve damage to brain microvasculature but the exact underlying cascade of events, including a potential role for haemostasis, has yet to be elucidated. Haemostatic defects (congenital or acquired) may contribute to an increased number and importance of CMBs. Congenital bleeding disorders such as haemophilia or von Willebrand disease (vWD), populations at high risk of ICH, are unique conditions that may give us further insights into a potential role of haemostatic defects in the pathophysiology of CMBs. CMBs might be the missing link between severe haemostatic defects, ICH risk and cognitive function.

We hypothesized that severe congenital haemostatic defects could contribute to an increased prevalence and number of CMBs, with an impact on cognition in adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, older than 18 years old, no upper age limit
* Adult patients with a severe congenital haemostatic defect

  * Severe or moderate congenital haemophilia A (or B) defined as <5 IU/dL (<5%) endogenous FVIII (FIX) activity at screening
  * Severe von Willebrand disease defined as VWF: Act ≤15IU/dL (<15%) at screening
* Ability of the participant to provide signed and dated informed consent

Exclusion Criteria:

* Contraindication for brain MRI
* HIV infection to avoid a bias towards severe multifactorial neurological complications
* Other known coagulation disorder(s) in addition to haemophilia or von Willebrand disease
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participation in this study (with the delivery of an information note) will be offered to all eligible patients during a follow-up visit related to haemophilia or Von Willebrand Disease within the Haemostasis-Transfusion Department of the Lille University Hospital.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The rate of patients with at least one CMB on 3-Tesla brain MRI (using specific sequences dedicated to the detection of CMBs). | Within 3 Months after inclusion

SECONDARY OUTCOMES:
Number and anatomical location (deep/lobar) of CMBs on 3-Tesla brain MRI | Within 3 Months after inclusion
Multi-domain cognitive performances assessed by standardized scales as follows | Within 3 Months after inclusion
  - MoCA
Multi-domain cognitive performances assessed by standardized scales as follows | Within 3 Months after inclusion
  Memory: The free and cued selective reminding test (FCSRT, French version) ; The Wechsler digit span task will be used to examine verbal short term and working memory.
Multi-domain cognitive performances assessed by standardized scales as follows | Within 3 Months after inclusion
  - Processing speed and attention: digit symbol coding subtest of WAIS 4; the Continuous Performance Test (third edition, CPT3).
Multi-domain cognitive performances assessed by standardized scales as follows | Within 3 Months after inclusion
  - Executive function: The categorical and literal fluency test and the Trail-Making Test (TMT).
Multi-domain cognitive performances assessed by standardized scales as follows | Within 3 Months after inclusion
  - Social cognition: MINI-SEA)
Multi-domain cognitive performances assessed by standardized scales as follows | Within 3 Months after inclusion
  - Depression: CES-D
Multi-domain cognitive performances assessed by standardized scales as follows | Within 3 Months after inclusion
  - Anxiety: HAM-A
Multi-domain cognitive performances assessed by standardized scales as follows | Within 3 Months after inclusion
  - Fatigue: The Chalder Fatigue Scale
Multi-domain cognitive performances assessed by standardized scales as follows | Within 3 Months after inclusion
  - Sleepiness and the impact of sleep disorders: The Epworth Sleepiness Scale

IPD SHARING:
Plan to Share IPD: No